CLINICAL TRIAL: NCT00645762
Title: Balloon REmodeling Antrostomy THErapy Study (BREATHE I)
Brief Title: Balloon REmodeling Antrostomy THErapy Study
Acronym: BREATHE I
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Entellus Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1156-001
Record Dates: First submitted 2008-03-20; First posted 2008-03-28 (Estimated); Results first posted 2013-07-29 (Estimated); Last update posted 2013-07-29 (Estimated); Status verified 2013-06

CONDITIONS: Sinusitis
Keywords: Chronic rhinosinusitis; Chronic sinusitis; Maxillary sinus; Anterior ethmoid sinus; Ethmoid infundibulum; Balloon dilation; Endoscopic visualization; Local anesthesia; Canine fossa; Less invasive
MeSH Terms: conditions — Sinusitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Balloon Dilation (Active Comparator): Balloon dilation with FinESS device
  Interventions: Device: RS-Series Rhinosinusitis Treatment System; Device: FinESS Balloon

INTERVENTIONS:
Device: RS-Series Rhinosinusitis Treatment System — Single arm
Device: FinESS Balloon

SUMMARY:
This study is designed to evaluate safety and effectiveness of a less invasive procedure to treat maxillary only, or maxillary and anterior ethmoid, chronic sinusitis. Additionally, this study will assess the feasibility of performing the procedure under local anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Subjects age 18 or older with chronic rhinosinusitis of the maxillary or maxillary and anterior ethmoid sinuses
* A CT scan taken after maximal medical therapy (e.g., local or systemic antibiotics, topical steroids, etc.) must show one of the following:

  1. Narrowing of the outflow tract of the maxillary sinus ostium or infundibulum with mucosal thickening of 2 mm or greater of the maxillary sinus antrum.
  2. Evidence of maxillary sinus air/liquid level.

Exclusion Criteria:

* Evidence of chronic posterior ethmoid, sphenoid or frontal sinusitis
* Inability to understand the study or a history of non-compliance with medical advice
* Unwilling or unable to sign Informed Consent Form (ICF)
* Currently enrolled in any other pre-approval investigational study (does not apply to long-term post-market studies)
* History of any cognitive or mental health status that would interfere with study participation
* Previous sinus surgery or intervention including sinuplasty
* Pregnant women
* Severe septal deviation causing obstruction of the ostiomeatal unit
* History of primary ciliary dysfunction
* Hemophilia
* Currently undergoing or in the past 6 months had undergone chemotherapy for cancer or radiation therapy in the head or neck region
* History of cystic fibrosis
* Known Sampter's Triad (aspirin sensitivity, asthma, sinonasal polyposis)
* Known sinonasal tumors or obstructive lesions
* History of mid facial fractures or orthognathic surgery (does not include nasal fracture)
* History of insulin dependent diabetes
* Not able to stop anti-coagulant (e.g., warfarin) until the International Normalized Ratio(INR) is below 1.5
* Not able to stop anti-platelet (e.g., clopidogrel, aspirin, etc.) for at least 14 days prior to study procedure
* Not able to stop any non-steroidal anti-inflammatory medications and homeopathic medications for at least 14 days prior to the study procedure
* Presence of nasal polyps that may interfere with the treatment procedure
* Presence of features consistent with sinus fungal disease on CT or physical examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2007-09; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Stankiewicz, MD, Principal Investigator — Loyola University Medical Center, Maywood, IL; Thomas Tami, MD, Principal Investigator — Cincinnati Sinus Institute, Cincinnati OH
Locations (13):
- United States (13):
  - Central California Ear, Nose and Throat Medical Group, Fresno, California
  - NorthShore University HealthSystem, Evanston, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - St. Cloud Ear, Nose & Throat - Head and Neck Clinic, Saint Cloud, Minnesota
  - Otolaryngology-Facial Plastic Surgery of Long Island P.C., Lake Success, New York
  - Charlotte Eye, Ear, Nose & Throat Associates, Charlotte, North Carolina
  - Midwest Ear, Nose, and Throat, Sioux Falls, South Dakota
  - Holston Medical Group, Kingsport, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Austin Ear, Nose & Throat Clinic, Austin, Texas
  - Texas Sinus Center, Boerne, Texas
  - San Antonio Ear, Nose, and Throat Research, San Antonio, Texas
  - Ear, Nose, Throat & Plastic Surgery Associates, PS, Auburn, Washington

REFERENCES:
- [Derived] Stankiewicz J, Tami T, Truitt T, Atkins J, Liepert D, Winegar B. Transantral, endoscopically guided balloon dilatation of the ostiomeatal complex for chronic rhinosinusitis under local anesthesia. Am J Rhinol Allergy. 2009 May-Jun;23(3):321-7. doi: 10.2500/ajra.2009.23.3274. Epub 2009 Jan 16. PMID 19419611

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrolled patients with chronic rhinosinusitis (CRS) from Ear, Nose Throat (ENT) physician practices.
Pre-assignment Details: All patients had transantral balloon dilation of the maxillary sinus ostium and ethmoid infundibulum with the FinESS Sinus System.
Groups:
- FinESS Sisnus System Balloon Dilation: Transantral balloon dilation ofthe maxillary sinuses with the FinESS Sinus System.
Period: Overall Study
Arm/Group | FinESS Sisnus System Balloon Dilation
Started | 71
Completed | 67
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Balloon Dilation
Number analyzed (Participants) | 71
Age Continuous [Mean (Standard Deviation); unit: years] | 47.3 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 26
Region of Enrollment [Number; unit: participants]
  United States | 71

OUTCOME MEASURES:

1. Primary Outcome: Incidences of Device-related or Procedure-related Complications
Time Frame: Through 12 months post-procedure
Population: Patients completing 12 month follow-up
Measure: Number; unit: participants
Groups:
- Treatment Group (ALL): FinESS Balloon Dilation
Arm/Group | Treatment Group (ALL)
Number analyzed (Participants) | 67
participants | 1 (0.98)

2. Primary Outcome: Patency of the Treated Area as Verified by CT Scan
Description: Post-procedure Patency was assessed using a CT scan 3 months post-procedure. The osteomeatal complex was assessed for patency by physicians.
Time Frame: Post-treatment at 3 months
Population: Analysis of ostia patency done per protocol
Measure: Number; unit: Ostia
Units Other Than Participants: Treated Maxillary Ostia
Arm/Group | FinESS Balloon Dilation
Number analyzed (Participants) | 71
Number analyzed (Treated Maxillary Ostia) | 117
Ostia | 106

3. Primary Outcome: Symptomatic Score Change- Sinonasal Outcome (SNOT) 20 Score Improvement
Description: Symptomatic change in SNOT 20 scores on a 5-point Likert scale where "0" = no problem to "5" = problem as bad as it can be were calculated. Baseline scores and 12 month post-procedure follow-up scores were calculated and compared. A score reduction of at least 0.8 (-0.8) from baseline to 12 months is considered statistically significant and clinically impactful.
Time Frame: Post-treatment through 12 months
Population: Score reduction in SNOT 20 Scale Scores. Baseline through 12 months post-procedure.
Measure: Number; unit: Scores on a scale
Groups:
- FinESS Balloon Arm: Subjects completing 12 month post-procedure follow-up
Arm/Group | FinESS Balloon Arm
Number analyzed (Participants) | 67
Scores on a scale | -1.8

ADVERSE EVENTS:
Time Frame: 12 months post-procedure
Arm/Group | Treatment Group (ALL)
Serious Adverse Events (participants affected / at risk) | 1/71
Other Adverse Events (participants affected / at risk) | 0/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group (ALL) (N=71)
Subcutaneous emphysema of the neck and upper chest (Skin and subcutaneous tissue disorders) | 1 (1) — Continuous positive airway pressure (CPAP) usage resumed same day as procedure.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days